CLINICAL TRIAL: NCT02328456
Title: A Randomized Controlled Trail to Determine the Impact of a SMS Reminder Associated With Free Eye Drops on Follow-up Adherence After Trabeculectomy Surgery in Rural China
Brief Title: Effect of SMS Reminder and Free Eye Drops on Follow-up Adherence After Trabeculectomy Surgery in Rural China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Congdon Nathan (Other)
Collaborators: Orbis (Other)
Responsible Party: Sponsor-Investigator, Congdon Nathan, vice directior,Blindness Prevention and Treatment Department, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ZOC-CREST-COMPLIANCE-GLAUCOMA
Record Dates: First submitted 2014-12-23; First posted 2014-12-31 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Glaucoma; Adherence
MeSH Terms: conditions — Glaucoma | interventions — Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS and free eye drops group (Other): the patient after trabeculectomy surgery in the SMS associated with free eye drops group will receive free eye drops and a SMS reminder message about the revisit time.
  Interventions: Other: SMS and free eye drops
- the control group (No Intervention): the patient after trabeculectomy surgery in the control group won't get any free eye drop and reminder message before the appointment.

INTERVENTIONS:
Other: SMS and free eye drops — The SMS reminder message will sent to the SMS associated with free eye drops group patients 1 week and 1 day before there appointment to remind them the exact time and address of the revisit appointment.The eye drops will be offered free to the the SMS associated with free eye drops group patients when they revisit on time.
  Arms: SMS and free eye drops group

SUMMARY:
The purpose of the study is to use a randomized controlled design to determine the impact of a SMS messaging associated with free eye drops intervention on the following outcomes among patients after trabeculectomy surgery in rural China.

DETAILED DESCRIPTION:
SMS message reminder is a system which can sent re-visit information to remind the patient about the revisit time and address. The investigators can use the SMS system to find out if it is a useful to reduce the not-attended rate of the revisit appointment among the rural patients.

ELIGIBILITY:
Inclusion Criteria:

* All the patients after trabeculectomy surgery in 4 cooperated rural hospitals

Exclusion Criteria:

* Both the patient and his/her caretakers don't have cellphone or the one who has cellphone but don't know how to use the SMS function.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Not-attended rate | up to 1 year
  Compare the SMS and free eye drops patient not-attend rate with the control group to show the impact of SMS reminder associated with free eye drops on the adherence with scheduled follow-up visit

SECONDARY OUTCOMES:
Knowledge and Attitudes about glaucoma, glaucoma surgery and importance of follow-up using a questionnaire | up to 1 year
  Using a questionnaire to compare Knowledge and Attitude between the SMS associated with free eye drops group and the control group
Additional factors potentially associated with post-operative follow-up using a patient questionnaire | up to 1 year
  Using a patient questionnaire to compare between the SMS associated with free eye drops group and the control group

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Congdon, MD,MPH, Study Director — China,Guangdong,Blindness Preventment and Treatment Department,Zhongshan Ophthalmic Center,510060
Locations (1):
- Blindness Preventment and Treatment Department, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang K, Jin L, Li L, Zeng S, Wei R, Li G, Man P, Congdon N. Interventions to Promote Follow-up After Trabeculectomy Surgery in Rural Southern China: A Randomized Clinical Trial. JAMA Ophthalmol. 2016 Oct 1;134(10):1135-1141. doi: 10.1001/jamaophthalmol.2016.2819. PMID 27541442